CLINICAL TRIAL: NCT02134496
Title: PACU Discharge Without Motorfunction Assessment After Spinal Anaesthesia for Total Hip or Knee Arthroplasty - a Multicenter Randomized Controlled Trial
Brief Title: PACU Discharge Without Motorfunction Assessment After Spinal Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Eske Kvanner Aasvang, M.D. DMSci, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-1-2014-012
Record Dates: First submitted 2014-04-28; First posted 2014-05-09 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Osteoarthritis Susceptibility 3
Keywords: hip; knee; arthroplasty; spinal; anesthesia
MeSH Terms: interventions — Recovery Room

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- no assessment of motorfunction in PACU (No Intervention): no assessment of motorfunction after spinal anesthesia in PACU
- motorfunction assessment in PACU (Active Comparator): Assesment of motorfunction after spinal anesthesia
  Interventions: Procedure: assessment of motorfunction in PACU

INTERVENTIONS:
Procedure: assessment of motorfunction in PACU — assessment of motorfunction in PACU after spinal anesthesia
  Arms: motorfunction assessment in PACU

SUMMARY:
The study investigates the safety of discharge from the Post-Anesthesia Care Unit (PACU) without assessment of motorfunction after spinal anesthesia for total hip- or knee replacement. This is an randomized controlled trial between two groups with assessment of normal (Aldrete) PACU discharge criteria with or without assessment of the motorfunction. The study hypothesis is that it is safe to be discharged from the PACU to a ward without assessment of motor function.

The main outcome is length of hospial stay (LOS) in days and re-admission within the first 30 days after surgery .

Secondary outcomes include adverse events up to 24 hours after surgery, and minuttes spent in the PACU after surgery.

Participants will be monitores for adverse events for the first 24 hours after surgery and reported. The total number of minuttes spent in the PACU will be recorded and reported.

DETAILED DESCRIPTION:
A novel analysis of the latest database version was performed 06.04.2015, showing that 86.7% of patients have LOS of less than 5 days and no re-admission within the first 30 days after discharge.

The study is designed as a non-inferiority study with a two-sided 5% significance level, 80% power and a non-inferiority level of 5%, resulting in 2 x 725 patients (1500 in total including drop-outs).

A 30-day re-admission period was chosen to detect complications that could be assumed to have occurred as a consequence of the potential earlier PACU discharge The study will also investigate Length of stay, incidence of failed anesthesia, and reason for stay in PACU after THA and TKA 24.11.2016 A substudy based upon the un-published data from the time in PACU will be performed to analyse factors related to adverse events occuring during the PACU stay, and description of specific organdysfunction based upon the recordings from the modifed Aldrete discharge criteria.

Preoperative demographic data are collected from charts and the Lundbeck Centre for Fast-track Hip and Knee Replacement database, (LCDB), intraoperative data from anesthesia charts.

A logistic regression analysis will be performed with the YES/NO outcome of moderate/severe adverse PACU events at any time during PACU stay, and pre- and intr operatie variables.

ELIGIBILITY:
Inclusion Criteria:

* age 18 yr or more
* primary unilateral total hip or knee arthroplasty
* spinal anesthesia

Exclusion Criteria:

* intraoperative conversion to general anesthesia
* intraoperative bleeding exceeding 750 ml.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1511 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Lenght of stay (in days) or 30 day readmissions | 30 days
  The main outcome is a compund measure of the duration of hospitalization after operation )measured in days, and named Length of Stay LOS) adn/or re-admission within the first 30 days after discharge.

SECONDARY OUTCOMES:
Adverse events | 24 hours postooperatively
  Any event that results in a physicians assessment of the patient, not including regular rounds during the first 24 hours after surgery.

OTHER OUTCOMES:
Time to discharge from PACU | 12 hours
  Time from arrival to discharge i PACU measured in minuttes
Discharge readiness before leaving the operating theater | 1 hour
  How many patients fulfilled the PACU discahrge criteria at the time they were leaving the operating theater
Failed spinal anesthesia. | 6 hours.
  Incidence and related factors to failed spinal anesthesia (ie. conversion to generel anesthesia)
Prediction of PACU complications | 0-7 hours
  Factors related to, and incidence of, moderate/severe complications i PACU

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Kehlet, Professor, Study Chair — Rigshospitalet, Denmark; Eske K Aasvang, M.D., DMSci, Principal Investigator — Rigshospitalet, Denmark
Locations (5):
- Denmark (5):
  - Gentofte Hospital, Gentofte Municipality, International
  - Vejle Sygehus, Vejle, International
  - Farsø Sygehus, Farsø
  - Holstebro Sygehus, Holstebro
  - Viborg Hospital, Viborg

REFERENCES:
- [Derived] Aasvang EK, Laursen MB, Madsen J, Kroigaard M, Solgaard S, Kjaersgaard-Andersen P, Mandoe H, Hansen TB, Nielsen JU, Krarup N, Skott AE, Kehlet H. Incidence and related factors for intraoperative failed spinal anaesthesia for lower limb arthroplasty. Acta Anaesthesiol Scand. 2018 Aug;62(7):993-1000. doi: 10.1111/aas.13118. Epub 2018 Mar 26. PMID 29578248